CLINICAL TRIAL: NCT02750553
Title: A Phase 1, Randomized, Placebo-controlled, Single & Multiple Dose Escalation Study to Investigate Safety, Pharmacokinetics, and Pharmacodynamics of SHR0534 in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0534-Ia
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
MeSH Terms: interventions — SHR0534

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Pre-test (Experimental): Three healthy male subjects were randomized in 2:1 ratio to receive single and then multiple (14 days) oral dose of 5 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 1 (Experimental): Eight healthy subjects were randomized in 3:1 ratio to receive single and then multiple (14 days) oral dose of 5 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 2 (Experimental): Ten healthy subjects were randomized in 4:1 ratio to receive single and then multiple (14 days) oral dose of 10 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 3 (Experimental): Ten healthy subjects were randomized in 4:1 ratio to receive single and then multiple (14 days) oral dose of 25 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 4 (Experimental): Ten healthy subjects were randomized in 4:1 ratio to receive single and then multiple (14 days) oral dose of 50 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 5 (Experimental): Ten healthy subjects were randomized in 4:1 ratio to receive single and then multiple (14 days) oral dose of 100 mg SHR0534 or matching placebo.
  Interventions: Drug: SHR0534; Drug: Placebo

INTERVENTIONS:
Drug: SHR0534
Drug: Placebo

SUMMARY:
This is a randomized, placebo-controlled, single & multiple dose escalation study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR0534. The study will be conducted with starting dose of 5 mg followed by dose escalation groups up to 100 mg. Healthy Chinese subjects will be randomized in each cohort to receive the study drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Must have a BMI between 18 to 24.9 kg/m2, inclusive;
* Clinical laboratory tests (i.e.blood chemistries, and urinalysis) must be within the normal reference range or clinically acceptable as determined by the investigator;
* Subjects must be free of any clinically significant diseases based on medical history , physical examination and/or the investigator's judgment;
* Winthout bad habits, including smoking, drinking and others;
* Negative in Urine or serum pregnancy test for woman, female subject of childbearing potential and male subject must be willing to use an acceptable method of birth control for the duration of the study and continuing 90 days after discontinuing treatment with the investigational ;
* Subject must be able to understand the information associated with the study, and are willing to provide written informed consent.

Exclusion Criteria:

* Clinically relevant abnormalities of physical examination, laboratory values, vital signs or ECG findings at the screening, as judged by the Investigator;
* History of surgery or major trauma within 12 weeks of study entry, or surgery planned during the study;
* History of hypersensitivity to SHR0534 or its components;
* Any condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, or a history of severe unconsciousness hypoglycemia judged by researchers;
* History of liver disease. Those with Alanine aminotransferase (ALT) or Aspertate aminotransferase (AST)>1.5 times upper limit of normal must be excluded;
* Severe infection, trauma or major surgery 4 weeks before screening;
* Congestive heart failure and other serious heart and lung diseases that need medication;
* Have a positive test at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb);
* Positive in nicotine screening test, or cannot refrain from smoking;
* Urine drug screen test positive for ethanol, cocaine, tetrahydrocannabinol (THC), barbiturates, amphetamines, benzodiazepines, or opiates;
* Subject who cannot refrain from smoking, eating and/or drinking containing xanthine/caffeine, or strenuous exercise, or others that affect drug absorption, distribution, metabolism and excretion within 2 days before the study drug administration;
* Have used any drugs or substances (including herbal supplements) known to inhibit or induce cytochrome (CYP) P450 enzymes including CYP3A4, CYP2C8 and CYP2C9 within 28 days prior to the first dose and throughout the study;
* Use of any prescription drugs and Chinese herbal medicines within 4 weeks before randomization, or use of non prescription drugs and food supplements (vitamins, etc.) within 2 weeks before randomization;
* Participated any drug clinical trials within 3 months, or had blood donation/loss ≥500 mL within 4 weeks before randomization;
* Female subject of childbearing potential who does not use an acceptable method of birth control, is pregnant or planning a pregnancy, or breastfeeding, or male subject who does not use an acceptable method of birth control, within six months before randomization;
* Subject who is unsuitable for inclusion in the study in the opinion of he investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From baseline up to 8 days after last treatment (Day 31)

SECONDARY OUTCOMES:
Area under the plasma or urine concentration curve after single or the last multiple oral dose (AUC) | From time 0 to 168 hours for single dose, and from time 0 to 192 hours after the last dose
Peak plasma concentration (Cmax) after single or the last multiple oral dose | From time 0 to 168 hours for single dose, and from time 0 to 192 hours after the last dose
Terminal elimination halflife (t½) for SHR0534 after single or the last multiple oral dose | From time 0 to 168 hours for single dose, and from time 0 to 192 hours after the last dose
Changes in the concentrations of blood glucose and insulin after single or multiple oral dose | From baseline up to 24 hours after last treatment (Day 24)

IPD SHARING:
Plan to Share IPD: No